CLINICAL TRIAL: NCT02309021
Title: PHAST: Influence of Exercise Training on Substance Use, Substance Craving, Quality of Life, Mental Health, Sleep, and Physical Health in Patients Suffering From Opiate Dependence While Under Substitution Therapy
Brief Title: PHAST: Physical Activity in Substitution Therapy
Acronym: PHAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Psychiatric Hospital of the University of Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UHospitalSwitz
Record Dates: First submitted 2014-11-27; First posted 2014-12-05 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Substance-related Disorders
Keywords: craving
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sport Group (Other): Participants randomised to the exercise condition will receive 12 weeks of physical exercise training. Once they have been assigned to this group, they will be informed about the training programme and its content. Training will be carried out in groups (two groups of ten or four groups of five, depending on scheduling, sport preferences, available materials) to ensure that individual attention can be paid to each participant.
  Interventions: Other: Sport
- Control Group (Other): The control group will not receive any exercise training. In order to control, as far as possible, for the potentially therapeutic effects of extra contact time with investigators, and the potentially motivational elements of participation in an intervention, the C group will have equal contact time with an investigator and participate in a leisure program without physical activity component. This time will be filled with group mealtimes, games, films, painting, handcrafts, stretching or relaxation exercises.
  Interventions: Other: Non-sport activities

INTERVENTIONS:
Other: Sport
  Arms: Sport Group
Other: Non-sport activities
  Arms: Control Group

SUMMARY:
The aim is to examine the effect of exercise (EX) training on individuals currently receiving ST - either opiate replacement therapy (ORT) or heroin-assisted treatment (HAT) - for their opiate dependence. Main outcome variables will be: cardiovascular fitness; consumption of substances (e.g. "street heroin", cocaine, cannabis, alcohol, cigarettes) other than prescribed ST or other prescribed medications; substance craving; blood pressure; lung function; resting pulse; social interaction; self-control capacity; objective and subjective sleep; cortisol levels; quality adjusted life years (QALYs); depression; mood. Covariates are current substitution dose and psychiatric diagnoses.

DETAILED DESCRIPTION:
The investigators aim is to carry out a randomized controlled trial comparing exercise training group and a control group of patients receiving substitution therapy (ST). The specific goals of the study are:

1. To understand the exercise preferences, barriers to participation, motivation, experiences and attitudes regarding exercise training in patients under ST.
2. To examine whether a 12-week exercise programme affects the mental health, subjective and objective sleep, quality of life, self-control capacity, substance craving, hair cortisol levels, secondary consumption, cardiovascular fitness, blood pressure, lung function, resting pulse, and social interaction in patients receiving ST.
3. To compare the effects of the EX and control conditions on the above-mentioned outcome variables.
4. To examine to what degree the covariates of heroin substitution dose and psychiatric comorbidities affect outcome variables.
5. To explore to what extent objective variables (cardiovascular fitness, pulse, blood pressure, lung function, cortisol, objective sleep-EEG-parameters) and subjective-psychological dimensions (subjective sleep, social interaction, symptoms of depression and anxiety, self-control, substance craving) are interrelated.

ELIGIBILITY:
Inclusion Criteria:

Patient at the Ambulanter Dienst Sucht or Janus clinics in Basel Town (BS); currently under substitution therapy

Exclusion Criteria:

Declared unfit to participate by clinic personnel due to physical disability or severe psychological disturbance or cognitive impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Craving measured by the Brief Substance Craving Scale (translated) | 6 months
  Craving will be measured by the Brief Substance Craving Scale (translated)
Secondary substance consumption assessed using the Time Line Follow Back method | 6 months
  This will be assessed using the Time Line Follow Back method

SECONDARY OUTCOMES:
Depression assessed using the Allgemeine Depressionskala ( Depression Scale) | 6 months
  Depression will be assessed using the Allgemeine Depressionskala ( Depression Scale)
Self control measured using the Short Self Control Scale (translated) | 6 months
  This will be measured using the Short Self Control Scale (translated)
Subjective sleep measured using the Insomnia Severity Index (translated) | 6 months
  This will be measured using the Insomnia Severity Index (translated)
Physical activity level measured using the International Physical Activity Questionnaire | 6 months
  This will be measured using the International Physical Activity Questionnaire
Perceived Stress measured using the Perceived Stress Scale (translated) | 6 months
  Will be measured using the Perceived Stress Scale (translated)
Quality adjusted life years assessed using the Short Form (SF)36 questionnaire | 6 months
  This will be assessed using the Short Form (SF)36 questionnaire
Blood pressure measured using a digital sphygmomanometer | 6 months
  This will be measured using a digital sphygmomanometer
Lung function measured with a Spirobank Spirometer | 6 months
  Lung function will be measured with a Spirobank Spirometer
Hand grip strength assessed using a Hydraulic Hand Dynamometer. | 6 months
  This will be assessed using a Hydraulic Hand Dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Flora Colledge, PhD, Principal Investigator — Department for Sport, Exercise and Health
Locations (1):
- Department for Sport, Exercise and Health, Basel, Switzerland